CLINICAL TRIAL: NCT04199988
Title: Reliability of Posterior Shoulder Endurance Test in Overhead Athletes and Comparison of Athletes With and Without Shoulder Pain
Brief Title: Reliability of Posterior Shoulder Endurance Test in Overhead Athletes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Damla Karabay, Research assistant, Dokuz Eylul University
Other Study IDs: 4950-GOA
Record Dates: First submitted 2019-12-11; First posted 2019-12-16 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Shoulder Pain; Healthy
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Athletes with shoulder pain: Overhead athletes with shoulder pain
  Interventions: Diagnostic Test: Posterior Shoulder Endurance Test
- Athletes without shoulder pain: Overhead athletes without shoulder pain
  Interventions: Diagnostic Test: Posterior Shoulder Endurance Test

INTERVENTIONS:
Diagnostic Test: Posterior Shoulder Endurance Test — Isometric posterior shoulder endurance test: In the prone position, the athlete's shoulder will be placed at horizontal abduction, and the time for maintaining this position will be recorded.
  Isotonic shoulder endurance test: In the prone position, the athlete's shoulder will be placed at horizontal abduction and asked to perform horizontal adduction-abduction, and the athlete will horizontally abducted-adducted his/her arm to 90 degrees at a cadence of 30 beats per minute. The number of repetitions will be recorded.

SUMMARY:
The purpose of this study was to investigate the reliability of posterior shoulder endurance test in overhead athletes and to compare the endurance of posterior shoulder muscles between athletes with and without shoulder pain.

DETAILED DESCRIPTION:
A total of 40 overhead athletes, 20 with shoulder pain and 20 with no shoulder pain, will be included in the study. Shoulder endurance will be measured as isometric and isotonic on both arms of athletes using the posterior shoulder endurance test. The measurements will be repeated after 3-7 days, and the test-retest reliability of the isotonic and isometric posterior shoulder endurance test will be investigated.

ELIGIBILITY:
Inclusion Criteria:

For all athletes:

* Being between the ages of 13-24,
* Participating to overhead sports (tennis, volleyball, handball, etc.),
* Training at least 2-3 hours a week,
* Active participation in training and competitions,
* To be able to complete all assessments in the study,

For athletes with shoulder pain:

* Shoulder pain is 3/10 or more in the Visual Analogue Scale.

For Athletes without shoulder pain:

* No shoulder pain (0/10 according to Visual Analog Scale)
* No history of a shoulder injury and/or shoulder symptoms requiring treatment for the past 1 year.
* Having 90/100 or higher results in Kerlan-Jobe Orthopedic Clinical Shoulder & Elbow Score

Exclusion Criteria:

* Bilateral shoulder pain,
* Upper extremity fracture history,
* Surgical history of shoulder, cervical and thoracic region,
* Diagnosis of musculoskeletal disease in the cervical region, elbow, and wrist,
* Neck and shoulder pain with active/passive cervical spine movement,
* Frozen shoulder,
* Multidirectional joint hypermobility,
* Having a systemic musculoskeletal disease,
* Diagnosis of chest deformity and scoliosis.

Ages: 13 Years to 24 Years | Sex: All
Age Groups: Child, Adult
Study Population: Overhead athletes with and without shoulder pain
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Isometric Posterior Shoulder Endurance Test | Measurements will be performed in two sessions (3 to 7 days)
  Isometric
Isotonic Posterior Shoulder Endurance Test | Measurements will be performed in two sessions (3 to 7 days)
  Isotonic

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi Sevi YESİLYAPRAK, PhD, Principal Investigator — Dokuz Eylul University; Birsu TOPÇUGİL KIRIK, MD, Study Chair — Dokuz Eylul University; Oğuz YÜKSEL, MD, Study Chair — Dokuz Eylul University; Oğuzcan GÖKÇAY, MD, Study Chair — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Sports Medicine department, Balçova, İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No